CLINICAL TRIAL: NCT04040608
Title: Influence of Screen Sizes on Responses to Visual Analog Scales of Stress
Acronym: SIVAStress
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Institut de Médecine du Travail (Unknown); UMR CNRS 6024, LaPSCo (Unknown)
Responsible Party: Sponsor
Other Study IDs: RNI 2018 DUTHEIL 3; 2018-A03280-55 (Other: 2018-A03280-55)
Record Dates: First submitted 2019-07-26; First posted 2019-07-31 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Volunteers
Keywords: visual analog scale; stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental group: differences in responses to visual analog scales depending on screen sizes
  Interventions: Other: Influence of screen sizes on responses to visual analog scales of stress

INTERVENTIONS:
Other: Influence of screen sizes on responses to visual analog scales of stress — An open questionnaire will be created by the Clinical Research Direction. The questionnaire will be opened by the examinator who will fulfill the anonymized identification of participants and the type of screens. In a dedicated room at the LaPSCo, the participants will answer the same VAS on four different sizes/types of screens (24-inch screen, laptop, tablet, smartphone) and on paper. Saliva will be collected after answering questionnaires. Heart rate variability and skin conductance will be measured with the use of a wrist watch during 15 minutes, from the entrance in the room to the completion of questionnaires.
  The participant will undergo the same examination within a week (15 minutes).

SUMMARY:
Visual analog scales (VAS) are one of the most common tools used in questionnaires. VAS are validated for pain and stress for example on a horizontal, non-calibrated line of 100 mm, ranging from very low (0) to very high (100). Nowadays, most VAS are used on questionnaires on internet. However, the influence of screen sizes on responses to visual analog scales were never studied.

DETAILED DESCRIPTION:
Visual analog scales (VAS) are one of the most common tools used in questionnaires. VAS are validated for pain and stress for example on a horizontal, non-calibrated line of 100 mm, ranging from very low (0) to very high (100). Nowadays, most VAS are used on questionnaires on internet. However, the influence of screen sizes on responses to visual analog scales were never studied.

Primary objective is to study the influence of screen sizes on response responses to visual analog scales.

Secondary objectives are to assess:

* the variability of responses depending on screen sizes within a week
* the influence of perception of work and addiction to work on the variability depending on screen sizes
* relationships with biomarkers of stress : salivary DHEAS, heart rate variability and skin conductance

An open questionnaire will be created by the Clinical Research Direction. The questionnaire will be opened by the examinator who will fulfill the anonymized identification of participants and the type of screens. In a dedicated room at the LaPSCo, the participants will answer the same VAS on four different sizes/types of screens (24-inch screen, laptop, tablet, smartphone) and on paper. Saliva will be collected after answering questionnaires. Heart rate variability and skin conductance will be measured with the use of a wrist watch during 15 minutes, from the entrance in the room to the completion of questionnaires.

The participant will undergo the same examination within a week (15 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Adult persons

Exclusion Criteria:

* Refusal to participate in the study
* Unable to answer basic questions (difficulties understanding, cognitive disorders…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healhy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale to assess the perceived stress | day 0
  Visual analog scale to assess the perceived stress on a horizontal, non-calibrated line of 100 mm, ranging from very low (0) to very high (100)
Visual analog scale to assess the perceived stress | day 7
  Visual analog scale to assess the perceived stress on a horizontal, non-calibrated line of 100 mm, ranging from very low (0) to very high (100)

SECONDARY OUTCOMES:
Visual analog scale to assess anxiety | day 0, day 7
  Visual analog scale to assess anxiety on a horizontal, non-calibrated line of 100 mm, ranging from very low (0) to very high (100)
Visual analog scale to assess sleep quality | day 0, day 7
  Visual analog scale to assess sleep quality on a horizontal, non-calibrated line of 100 mm, ranging from very low (0) to very high (100)
Visual analog scale to assess fatigue | day 0, day 7
  Visual analog scale to assess fatigue on a horizontal, non-calibrated line of 100 mm, ranging from very low (0) to very high (100)
Job Demand-Control-Support (JDSC) questionnaire of Karasek | day 0, day 7
  The Job Demand-Control-Support (JDSC) questionnaire of Karasek assessed job demands, job control and social support through 26 items.
The Effort-Reward Imbalance Questionnaire (ERI) | day 0, day 7
  The Effort-Reward Imbalance Questionnaire (ERI) is a self-administrated test assessing psychological distress and health problems that may occur when there is an imbalance between the efforts required by the work and the rewards received.
The Work Addiction Risk Test (WART) | day 0, day 7
  The Work Addiction Risk Test (WART) was developed by Robinson et al. from symptoms reported by clinicians caring for patients with work addiction
Hospital Anxiety and Depression (HAD) Scale | day 0, day 7
  Hospital Anxiety and Depression (HAD) Scale is a self-reported questionnaire composed of 14 items with a 4-point Likert scale assessing anxiety (7 items) and/or depressive (7 items) symptoms
The Maslach Burn-out Inventory (MBI) | day 0, day 7
  The Maslach Burn-out Inventory (MBI) is composed of 22 items designed to assess the three components of the burn-out syndrome: emotional exhaustion (9 items), depersonalization (5 items) and reduced personal accomplishment (8 items)
Heart rate variability | day 0, day 7
  Heart rate variability and skin conductance will be measured with the use of the wristband Empatica E4, Italy
: skin conductance | day 0, day 7
  Heart rate variability and skin conductance will be measured with the use of the wristband Empatica E4, Italy
Salivary DHEAS | day 0, day 7
  Salivary DHEAS is a biomarker of chronic stress, with a long half-life of 16 hours

CONTACTS AND LOCATIONS:
Overall Officials: frédéric Dutheil, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No